CLINICAL TRIAL: NCT01841710
Title: Genetic Variability in Taste Perception
Status: Completed | Type: Observational
Sponsor: Monell Chemical Senses Center (Other)
Collaborators: Children's Hospital of Philadelphia (Other); University of Pennsylvania (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Julie A. Mennella, Member, Monell Chemical Senses Center
Other Study IDs: 816980; R01DC011287 (NIH)
Record Dates: First submitted 2013-04-24; First posted 2013-04-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: Bitter Taste; Pediatric Medications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women

SUMMARY:
This proposal describes a pilot study aimed at determining whether genetic variations in taste receptors determine differential taste tolerability of pediatric medications.

DETAILED DESCRIPTION:
This is a cross-sectional call-back study of taste perception and the relationship between taste perception and taste receptor genotype.

ELIGIBILITY:
Inclusion Criteria:

* Adult females who were previously enrolled in Efficacy of Bitter Blockers on Taste Acceptance in Pediatric Populations Study (Protocol #809789)

Exclusion Criteria:

* Women who are pregnant
* Women on drugs with potential serious adverse effects that are mediated through cytochrome P450.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One hundred women who were previously enrolled in the study entitled "Efficacy of Bitter Blockers on Taste Acceptance in Pediatric Populations," Protocol #809789; will be recruited for the current study
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Psychophysical data for taste solutions | 1-2 hours
  Primary outcome variables are intensity ratings of pediatric medications as well as a variety of generally recognized as safe bitter and non-bitter compounds.

SECONDARY OUTCOMES:
Maternal practices and perceptions of medication use | 1-2 hours
  Secondary outcome variables include questions related to maternal practices and perceptions of medication use and compliance of their children.

CONTACTS AND LOCATIONS:
Overall Officials: Julie A. Mennella, PhD, Principal Investigator — Monell Chemical Senses Center; Elizabeth Lowenthal, MD MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Monell Chemical Senses Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Mennella JA, Mathew PS, Lowenthal ED. Use of Adult Sensory Panel to Study Individual Differences in the Palatability of a Pediatric HIV Treatment Drug. Clin Ther. 2017 Oct;39(10):2038-2048. doi: 10.1016/j.clinthera.2017.08.012. Epub 2017 Sep 18. PMID 28923290